CLINICAL TRIAL: NCT06285500
Title: UNIQUE: Umbrella N-of-1 Tumor Trials - Umbrella Protocol for Oncology Single Patient Protocols
Brief Title: Umbrella Study for Single Patient Treatments in Oncology
Acronym: UNIQUE
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UNIQUE; 23-5095 (Other: University Health Network)
Record Dates: First submitted 2024-02-07; First posted 2024-02-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer; Rare Diseases
Keywords: single patient protocols
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: N-of-1 treatment with marketed drugs used on or off-label as per SOC.
  Interventions: Other: Patient-specific treatments
- Group 2: N-of-1 treatment with drugs accessed from SAP.
  Interventions: Other: Patient-specific treatments
- Group 3: N-of-1 treatment with non-marketed investigational agents.
  Interventions: Other: Patient-specific treatments

INTERVENTIONS:
Other: Patient-specific treatments — Treatment will be decided specifically for the patient based on biomarker test results.

SUMMARY:
The purpose of this study is to collect data for assessing the improvement of the overall response rate for the overall cohorts and the proportion of patients accessing precision targeted therapy.

DETAILED DESCRIPTION:
The UNIQUE umbrella protocol is an overarching framework to study precision medicine in patients with precise molecular data, who have exhausted all established treatment options and who are not eligible for any of the ongoing trials. Participants who have received/who may receive the following treatments may join the study and will be assigned to a study cohort (group):

* Group 1 - Health Canada approved/marketed drug(s) used on or off-label as per Standard of Care (SOC)
* Group 2 - Drugs accessed from Special Access Program (SAP)
* Group 3 - Non-marketed investigational agents

Under the UNIQUE framework, data from participants will be evaluated. The following data will be collected:

* Demographic data (for example: sex, race, month and year of birth)
* Medical history
* Cancer characteristics including biomarkers
* Treatment history
* response to treatment

ELIGIBILITY:
Inclusion Criteria & Exclusion Criteria:

Patient's existing genomic information from tumor molecular profiling will be discussed in the hospital expert molecular tumor board rounds consisting of representatives from specialist genomic profiling and medical oncology departments to decide N of 1 treatment for the patient. The discussion will surround the best next therapeutic option in the patient's cancer subtype with or without clear standard of care guidelines. Therefore, specific eligibility criteria aside from individual patient's medical history is not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have advanced and rare cancer with limited treatment options.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate for the overall cohorts and the number of patients accessing precision targeted therapy | 3 years

SECONDARY OUTCOMES:
Overall survival rate | 5 years
Progression-free survival | 5 years
Number of participants with adverse events as assessed by CTCAE v5.0 | 3 years
  For Groups 1 and 2: Only Grade 3 and above AEs/AESIs and SAEs that are related (possibly, probably or definitely) to the study drug.
  For Group 3: All SAEs (regardless of causality).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Dr., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No